CLINICAL TRIAL: NCT04141566
Title: Pseudo Continent Perineal Colostomy vs Permanent Left Iliac Colostomy After Abdominoperineal Resection for Ultra Low Rectal Adenocarcinoma: Comparaison of Out of Pocket Costs, Hospital Bills and Quality of Life
Brief Title: Pseudo Continent Perineal Colostomy vs Permanent Left Iliac Colostomy After Abdominoperineal Resection for Ultra Low Rectal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Collaborators: Institut National d'Oncologie Sidi Mohammed Ben Abdellah (Unknown)
Responsible Party: Principal Investigator, Amine Souadka, professor, Moroccan Society of Surgery
Other Study IDs: PCPC_PLIC
Record Dates: First submitted 2019-10-20; First posted 2019-10-28 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Rectal Neoplasms; Colostomy Stoma; Quality of Life
Keywords: Pseudocontinent perineal colostomy; Abdominoperineal resection; colostomy; Cost effectiveness; quality of life
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCPC: pseudocontinent perineal colostomy using shmidt technique for perineal reconstruction after abdominoperineal resection
  Interventions: Procedure: Perineal pseudocontinent colostomy
- PLIC: Permanenet left iliac colostomy , the standard technique after abdominoperineal resection and primary closure of the perineal wound
  Interventions: Procedure: Permanent left iliac colostomy

INTERVENTIONS:
Procedure: Perineal pseudocontinent colostomy — The procedure is performed in 2stages: as a usual APR starting by a laparoscopic approach esnsuring a complete mesorectal excision,then a perineal approach ensuring an extended excision of the entire internal and external sphincter complex, allowing the excision of the specimen.
  8to10cm of tof the colon is resected and harvested as a free graft, stripped of its meso and epiploics , then from its mucosa and placed in an antibiotic solution for 10min. This graft is wrapped snugly around the end of the colon 2-3 cm from its distal end for 1 and a half round. Absorbable 3.0 Sutures are taken to hold it in place. The end of the colon is brought out as a stoma in the perineum.
  Colonic irrigations are started from the third day according to the protocol previously reported. Patients and one of their family members are daily educated and assisted while performing colonic irrigations by specialized nurses.
  Groups: PCPC
Procedure: Permanent left iliac colostomy — After a usual laparoscopic APR, the perineal wound is closed and a permanent left iliac colostomy is performed
  Groups: PLIC

SUMMARY:
Aim of this study is to compare the cost-effectiveness and the quality of life in the 6 months following the surgery of a pseudo continent perineal colostomy (PCPC) and a permanent left iliac colostomy (PLIC) following an abdominoperineal resection (APR) for ultra low rectal cancer

DETAILED DESCRIPTION:
The surgical treatment of ultra low rectal adenocarcinoma has known great changes, yet the abdominoperineal resection (APR) is still indicated in over 20% of these cases.

A permanent left abdominal stoma is the standard salvage technique.

The pseudo continent perineal colostomy (PCPC) is an alternative technique especially in low income countries where the stoma bag and stoma care is not covered by health insurances.

Furthermore, this technique allows the conservation of body image, which is frequently requested by muslim patients whenever it is possible.

The aim of this study is to compare the cost effectiveness of both techniques as well as the quality of life of patients in the 6 first months following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years old or above
* Abdominoperineal resection for ultra low rectal cancer
* Creation of a definitive iliac colostomy or a pseudo continent perineal colostomy
* Patients willing to participate to this study (writting consent)

Exclusion Criteria:

-Patients unable to respond to the Quality Of Life questionnaires

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who underwent an abdominoperineal resection for ultra low rectal cancer with the creation of a definitive iliac colostomy or a pseudo continent perineal colostomy.
  The following informations will be collected : age, gender, type of stoma,operative aspects, postoperative morbidity according to Clavien score, out of pocket costs and out of pocket hospital bills, quality of life at 6 months after surgery according to EORTC 30 and CR29 QOL
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cost of management of both stoma types | 180 days from surgery
  defined by out of pocket costs during the first 6 months following the surgery in euros
Costs of hospital stay | 180 days from surgery
  defined as Out of pocket hospital bills in euros for all of the admission and the readmissions for surgical complication management
Globcal Quality of life of patients with PCPC and PLIC | 180 days from surgery
  using the EORTC C30 Quality Of Life questionnaires
Specific Quality of life of patients with PCPC and PLIC | 180 days from surgery
  using the EORTC CR29 Quality Of Life questionnaires

SECONDARY OUTCOMES:
90 day morbidity and mortality rate | 90 days from surgery
  defined by the Clavien Dindo rated from I to V at 90 post operative day.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institut of Oncology, Surgical oncology department, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Souadka A, Majbar MA, Amrani L, Souadka A. Perineal pseudocontinent colostomy for ultra-low rectal adenocarcinoma: the muscular graft as a pseudosphincter. Acta Chir Belg. 2016 Oct;116(5):278-281. doi: 10.1080/00015458.2016.1174020. Epub 2016 Jul 29. PMID 27472021
- [Background] Souadka A, Majbar MA, El Harroudi T, Benkabbou A, Souadka A. Perineal pseudocontinent colostomy is safe and efficient technique for perineal reconstruction after abdominoperineal resection for rectal adenocarcinoma. BMC Surg. 2015 Apr 10;15:40. doi: 10.1186/s12893-015-0027-z. PMID 25888423
- [Background] Souadka A, Majbar MA, Bougutab A, El Othmany A, Jalil A, Ahyoud FZ, El Malki HO, Souadka A. Risk factors of poor functional results at 1-year after pseudocontinent perineal colostomy for ultralow rectal adenocarcinoma. Dis Colon Rectum. 2013 Oct;56(10):1143-8. doi: 10.1097/DCR.0b013e31829f8cd5. PMID 24022531
- [Background] Dumont F, Souadka A, Goere D, Lasser P, Elias D. Impact of perineal pseudocontinent colostomy on perineal wound healing after abdominoperineal resection. J Surg Oncol. 2012 Jun 1;105(7):628-31. doi: 10.1002/jso.22105. Epub 2011 Sep 22. PMID 21953024
- [Background] Dumont F, Ayadi M, Goere D, Honore C, Elias D. Comparison of fecal continence and quality of life between intersphincteric resection and abdominoperineal resection plus perineal colostomy for ultra-low rectal cancer. J Surg Oncol. 2013 Sep;108(4):225-9. doi: 10.1002/jso.23379. Epub 2013 Jul 19. PMID 23868337